CLINICAL TRIAL: NCT02543580
Title: Transcutaneous Electrical Acupoint Stimulation Decreases Remifentanil Consumption and Postoperative Pain in Patients Undergoing Radical Mastectomy: Dual Acupoints Versus Single Acupoint in a Prospective Randomized Controlled Trial
Brief Title: TEAS-induced Analgesia: Dual vs Single Acupoints
Acronym: TADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Xijing Hospital (Other)
Responsible Party: Principal Investigator, wangqiang, Professor, Xijing Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: xijingmazui24
Record Dates: First submitted 2014-12-30; First posted 2015-09-07 (Estimated); Last update posted 2018-06-07 (Actual); Status verified 2018-06

CONDITIONS: Postoperative; Acute Pain; Chronic Pain
Keywords: mastectomy; transcutaneous electrical acupoint stimulation; acute pain; chronic pain
MeSH Terms: conditions — Acute Pain; Chronic Pain

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: For all patients, electrodes were placed at the bilateral PC6 and RN17 and connected to the Hwato Electric Acupuncture Treatment Instrument. No patients in the study had previous experience of undergoing transcutaneous electrical stimulation treatment. Patients were told that they might or might not feel the electrical stimulation. Interventions were performed by a designated investigator who was not involved in the anaesthesia or the follow-up. The stimulator was placed in an opaque box to blind the surgical team and the anaesthetists to the group allocation.
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- single acupoint (Experimental): transcutaneous electric acupoint stimulation is given at bilateral neiguan or 30min before anesthesia induction
  Interventions: Other: transcutaneous electric acupoint stimulation
- double acupoints (Experimental): transcutaneous electric acupoint stimulation is given at Danzhong and bilateral neiguan or 30min before anesthesia induction
  Interventions: Other: transcutaneous electric acupoint stimulation
- sham electroacupuncture (Experimental): electrode attached but no stimulation
  Interventions: Other: electrode attached but no stimulation

INTERVENTIONS:
Other: transcutaneous electric acupoint stimulation — electrodes are attached o the skin and electric stimulation is given
  Arms: double acupoints; single acupoint
Other: electrode attached but no stimulation — electrodes are attached o the skin but no stimulation is given
  Arms: sham electroacupuncture

SUMMARY:
The purpose of this study is to evaluate the effects of transcutaneous electric acupoint stimulation(TEAS) at single acupoint or dual acupoints on opioid consumption and postoperative pain in patients undergoing radical mastectomy

ELIGIBILITY:
Inclusion Criteria:

* patients aged from 18 to 65 yrs
* body mass index (BMI) of 18 to 30 kg/m2
* elective radical mastectomy under general anesthesia

Exclusion Criteria:

* contradictions to electric stimulation
* difficulties in communication
* histories of general anesthesia, drug or alcohol abuse or addiction
* cardiac dysfunction or severe hypertension, confirmed hepatic dysfunction and renal impairment
* participants recruited into other clinical trials during last three months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 153 (Actual)
Dates: Start 2015-07 (Actual); Primary Completion 2015-12 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
dose of remifentanil during anesthesia | from start of anesthesia to extubation, on average 2 hours

SECONDARY OUTCOMES:
time to recall | from end of remifentanil infusion to patient response to verbal command,approximately 10 minutes on average
  patient response to verbal command
time to extubation | from end of remifentanil infusion to extubation,approximately 10 minutes on average
incidence of respiratory depression during recovery | from extubation to discharge from post anesthesia care unit, approximately 40 minutes on average
incidence of nausea and vomiting during recovery | from extubation to discharge from post anesthesia care unit, approximately 40 minutes on average
visual analogue scale during recovery | from arriving to discharge from post anesthesia care unit, approximately 30 minutes on average
visual analogue scale at 24 hour after surgery | from end of surgery to 24 hours after surgery, totally 24 hours
pain score at 3 months after surgery | from discharge from hospital to 3 months after surgery, approximately 3 months
pain score at 6 months after surgery | from discharge from hospital to 6 months after surgery, approximately 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Lize Xiong, MD, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China